CLINICAL TRIAL: NCT01234233
Title: Effects of Preoperative Warming of Patients on Postoperative Hypothermia and Shivering.
Acronym: THER4-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, PD Dr. Jan Hoecker, PD Dr. Jan Höcker, University Hospital Schleswig-Holstein
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: THER-JH
Record Dates: First submitted 2010-09-09; First posted 2010-11-04 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Hypothermia
Keywords: hypothermia, accidental; prewarming; body temperature monitoring; preoperative warming; sublingual temperature assessment; tympanic temperature assessment
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 (No Intervention): Control group - no intervention: no preoperative warming
- Group 2 - 10 min prewarming (Active Comparator): 10 min prewarming preoperatively
  Interventions: Procedure: duration of preoperative active warming
- Group 3 - 20 min prewarming (Active Comparator): 20 min prewarming preoperatively
  Interventions: Procedure: duration of preoperative active warming
- Group 4 - 30 min prewarming (Active Comparator): 30 min prewarming preoperatively
  Interventions: Procedure: duration of preoperative active warming

INTERVENTIONS:
Procedure: duration of preoperative active warming — duration of prewarming by "forced air warming"
  Arms: Group 2 - 10 min prewarming; Group 3 - 20 min prewarming; Group 4 - 30 min prewarming

SUMMARY:
The investigators want to evaluate the effect of prewarming on the rate of postoperative hypothermia and shivering and to compare sublingual versus tympanic temperature assessment during the perioperative period in patients.

Patients will be randomly assigned to 4 groups with different duration of prewarming. Body temperature will be recorded regularly by sublingual and tympanic (by thermocouple) measurement. Incidence of hypothermia (temp. < 36°C) and shivering will be assessed postoperatively.

DETAILED DESCRIPTION:
Inadvertent perioperative hypothermia causes many serious complications. Therefore, prevention from, detection and therapy of hypothermia is essential. The appropriate methods of temperature assessment are still under debate as well as the effect and necessary duration of active prewarming of patients to avoid postoperative hypothermia and shivering.

The aim of our study is to evaluate the effect of prewarming on the rate of postoperative hypothermia and shivering and to compare sublingual versus tympanic temperature assessment during the perioperative period in patients undergoing elective minor surgery.

The investigators plan to include patients scheduled for routine minor surgery of approximately 1h duration. Patients will be randomly assigned to 4 groups with different duration of active prewarming. Body temperature will be recorded regularly by sublingual and tympanic (by thermocouple) measurement. Incidence of hypothermia (temp. < 36°C) and shivering will be assessed postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for minor surgery (planned duration approximately <1h).
* Age 18-75yrs,
* ASA I-II physical status

Exclusion Criteria:

* Emergency surgery,
* pregnant patients,
* patients not able to give informed consent,
* duration of surgery >2h,
* necessary postoperative mechanical ventilation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2010-03; Primary Completion 2011-03 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Incidence of hypothermic (body temperature < 36°C) patients at postoperative arrival at postoperative care unit (PACU) | postoperative arrival at PACU (once)
  After surgery patients will be admitted to PACU. Body temperature will be evaluted here to study the number of hypothermic patients depended from duration of preoperative warming.Time frame for assessment of data: 5 min after postoperative arrival at PACU (one single measurement, duration: 30 sec).Afterwards patients will be observed for about 2h.

SECONDARY OUTCOMES:
Performance of sublingual vs. tympanic temperature assessment preoperatively in awake patients. | preoperatively (once) at arrival at PACU
  Sublingual and tympanic body temperature will be assessed simultaneously once at patients' preoperative arrival at PACU and compared to each other with analysis of correlation. This means that one sublingual and one tympanic temperature value will be measured to be compared to each other.Time frame for assessment of data: one single measurement immediately (1 min) after patients' arrival at PACU. Afterwards: observation of patients for about 2h.
Performance of sublingual vs. tympanic temperature assessment intraoperatively in anaesthetised patients. | intraoperatively (30 min after start of surgery), once
  Sublingual and tympanic body temperature will be assessed simultaneously (once) 30 min after start of surgery and compared to each other with analysis of correlation. This means that one sublingual and one tympanic temperature value will be measured to be compared to each other.Time frame for data assessment: 1 min after 30 min after start of surgery.Afterwards patients will be observed for about 3h.
Performance of sublingual vs. tympanic temperature assessment postoperatively in awake patients. | at postoperative arrival at PACU, once
  Sublingual and tympanic body temperature will be assessed simultaneously (once) at patients' postoperative arrival at PACU and compared to each other with analysis of correlation. This means that one sublingual and one tympanic temperature value will be measured to be compared to each other.Time frame for data assessment: 30 sec immediately after patients' arrival at PACU.

CONTACTS AND LOCATIONS:
Overall Officials: Markus Steinfath, M.D., Study Director — Dep. of Anaesthesiology, UK-SH, Campus Kiel; Ernst P Horn, M.D., Principal Investigator — Klinikum Pinnerberg, Pinneberg, Germany; Jan Höcker, M.D., Principal Investigator — Dep. of Anaesthesiology, UK-SH, Campus Kiel; Berthold Bein, M.D., Study Chair — Dep. of Anaesthesiology, UK-SH, Campus Kiel
Locations (2):
- Germany (2):
  - UK-SH, Campus Kiel, Kiel, Schleswig-Holstein
  - Klinikum Pinnerberg, Dep. of Anaesthesiology, Pinneberg, Schleswig-Holstein

REFERENCES:
- [Derived] Hocker J, Bein B, Bohm R, Steinfath M, Scholz J, Horn EP. Correlation, accuracy, precision and practicability of perioperative measurement of sublingual temperature in comparison with tympanic membrane temperature in awake and anaesthetised patients. Eur J Anaesthesiol. 2012 Feb;29(2):70-4. doi: 10.1097/EJA.0b013e32834cd6de. PMID 22037543